CLINICAL TRIAL: NCT06981962
Title: Effectiveness of Nursing Interventions on the Prevention of Pressure Ulcers Among Immobile Stroke Patients
Brief Title: Nursing Interventions for the Prevention of Pressure Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Halmat Authman Rasheed, Assist professor, Hawler Medical University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Nursing interventions
Record Dates: First submitted 2025-05-07; First posted 2025-05-21 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Pressure Ulcer Prevention
Keywords: Immobile patient; Stroke; Pressure ulcers; Incidence; Nursing Intervention
MeSH Terms: conditions — Stroke; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: When the program is delivered, two group of high risk patients for pressure ulcer ( Braden scale score ≤12) will be compared for the development of pressure ulcer. The group that receive the program (64 patients) will compare with group that do not receive program (64 Patients).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Case (Experimental): The case group will receive appropriate pressure ulcer prevention program
  Interventions: Other: Pressure ulcer prevention program
- Control (No Intervention): In this study the control group will not receive pressure ulcer prevention program

INTERVENTIONS:
Other: Pressure ulcer prevention program — Interventions will consist of proper positioning, frequent change of patients' posture to limit or decrease pressure over the skin, skincare, such as maintaining adequate hydration, keep skin clean, prevent excessive dryness of skin, prevent message over bony prominence, and control moisture.
  Arms: Case

SUMMARY:
this study is aimed to assess the effectiveness of nursing interventions on the prevention of pressure ulcers among immobile stroke patients

DETAILED DESCRIPTION:
Research question: Question 1: What is the effect of nursing educational interventional program on the prevention of pressure ulcers among immobile stroke patients.

The interventional program will be provided for the patients over a period of two days in the hospital, then the pressure ulcer prevention program will demonstrated by the researcher. The education and demonstration will consist of proper positioning, frequent change of patients' posture to limit or decrease pressure over the skin, skincare, such as maintaining adequate hydration, keep skin clean, prevent excessive dryness of skin, prevent message over bony prominence, and control moisture.

A manual in the form of booklet will be given to the patients and their family caregiver.

ELIGIBILITY:
Inclusion Criteria:

1. Both gender
2. Patients' age ≥ 18 years old.
3. Patients who

   1. are at highly risk for pressure ulcer development.
   2. Braden scale score ≤ 12
   3. Are able to communicate clearly
   4. Provide written informed consent
   5. Do not participate in another study and do not receive any information regarding pressure ulcer prevention.

Exclusion Criteria:

1. Patients who have different types of mental problems
2. Braden scale score > 12
3. Have history of previous pressure ulcer and are unable to respond to verbal commands.
4. Patients who work as a health care provider.
5. Patients with different stages of pressure ulcer.

   -

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Change the incidence of pressure ulcer | 3 weeks follow up after patients discharge
  Patients' skin will be assessed for the development of pressure ulcer. A patient who move from high and very high-risk Braden scale score (≤12) to stage one pressure ulcer and above is considered as the occurrence of pressure ulcer event.
  Braden scale is a pressure ulcer risk assessment tool which evaluates ulcer formation areas such as elbow, occipital, sacrum, back, and heel and areas of bony prominences. 6 is the lowest total subscale score and 23 is the highest total subscale score. The lower total subscale scores, the higher risk for the development of pressure ulcer'

CONTACTS AND LOCATIONS:
Locations (1):
- Hawler Medical University, Erbil, Kurdistan, Iraq

IPD SHARING:
Plan to Share IPD: No